CLINICAL TRIAL: NCT00163423
Title: Comparison of Ciclesonide (80 mcg Once Daily in the Evening) and Fluticasone Propionate (100 mcg Twice Daily) in Patients With Mild to Moderate Asthma
Brief Title: Efficacy of Ciclesonide Versus Fluticasone Propionate in Patients With Mild to Moderate Asthma (12 to 75 y) (BY9010/M1-142)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BY9010/M1-142
Record Dates: First submitted 2005-09-12; First posted 2005-09-14 (Estimated); Last update posted 2016-12-08 (Estimated); Status verified 2016-12

CONDITIONS: Asthma
Keywords: Asthma; Ciclesonide; Fluticasone propionate
MeSH Terms: conditions — Asthma | interventions — ciclesonide

INTERVENTIONS:
Drug: Ciclesonide

SUMMARY:
The aim of the study is to compare the efficacy of ciclesonide versus fluticasone propionate on lung function, time to first asthma exacerbation, asthma symptoms, use of rescue medication, and quality of life in patients with mild to moderate asthma. Ciclesonide will be inhaled at one dose level once daily; fluticasone propionate will be inhaled at one dose level twice daily. The study duration consists of a baseline period (2 to 4 weeks) and a treatment period (24 weeks). The study will provide further data on safety and tolerability of ciclesonide.

ELIGIBILITY:
Main Inclusion Criteria:

* Outpatients
* Written informed consent
* History of bronchial asthma for at least 6 months
* Good health with the exception of asthma
* Treated with inhaled steroids with a maximum daily constant dosage of 250 mcg fluticasone propionate or equivalent
* FEV1 80 - 105% of predicted

Main Exclusion Criteria:

* Concomitant severe diseases or diseases which are contraindications for the use of inhaled steroids
* COPD (i.e. chronic bronchitis or emphysema) and/or other relevant lung diseases causing alternating impairment in lung function
* Current smoking with more than 10 pack-years
* Previous smoking with more than 10 pack-years
* Use of systemic steroids 4 weeks (injectable depot steroids 6 weeks) before entry into the baseline period, or more than 2 times
* Pregnancy
* Intention to become pregnant during the course of the study
* Breast feeding
* Lack of safe contraception

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 480
Dates: Start 2004-11; Primary Completion 2006-01 (Actual); Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
FEV1
time to the first asthma exacerbation.

SECONDARY OUTCOMES:
FVC
asthma symptom score
use of rescue medication
AQLQ(S) and EQ-5D
percentage of days on which patients perceived asthma control
percentage of nocturnal awakening-free days
percentage of rescue medication-free days
percentage of asthma symptom-free days
physical examination
vital signs
standard laboratory work-up
adverse events
number of patients with local oropharyngeal adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca AstraZeneca, Study Director — AstraZeneca
Locations (46):
- Austria (6):
  - Altana Pharma/Nycomed, Gmünd
  - Altana Pharma/Nycomed, Linz
  - Altana Pharma/Nycomed, Neusiedl/See
  - Altana Pharma/Nycomed, Perg
  - Altana Pharma/Nycomed, Steyr
  - Altana Pharma/Nycomed, Wiener Neustadt
- Canada (13):
  - Altana Pharma/Nycomed, Brandon
  - Altana Pharma/Nycomed, Hamilton
  - Altana Pharma/Nycomed, London
  - Altana Pharma/Nycomed, Mississauga
  - Altana Pharma/Nycomed, Montreal
  - Altana Pharma/Nycomed, Montreal, Quebec
  - Altana Pharma/Nycomed, Ottawa
  - Altana Pharma/Nycomed, Québec
  - Altana Pharma/Nycomed, Sainte-Foy, Quebec
  - Altana Pharma/Nycomed, Sarnia
  - Altana Pharma/Nycomed, Ste-Foy PQ
  - Altana Pharma/Nycomed, Toronto
  - Altana Pharma/Nycomed, Woodstock
- Germany (8):
  - Altana Pharma/Nycomed, Geesthacht
  - Altana Pharma/Nycomed, Hanover
  - Altana Pharma/Nycomed, Heidelberg
  - Altana Pharma/Nycomed, Koblenz
  - Altana Pharma/Nycomed, Mainz
  - Altana Pharma/Nycomed, Marburg
  - Altana Pharma/Nycomed, Sinsheim
  - Altana Pharma/Nycomed, Witten
- Poland (7):
  - Altana Pharma/Nycomed, Bielsko-Biala
  - Altana Pharma/Nycomed, Gdansk
  - Altana Pharma/Nycomed, Lodz
  - Altana Pharma/Nycomed, Lubin
  - Altana Pharma/Nycomed, Lublin
  - Altana Pharma/Nycomed, Wałbrzych
  - Altana Pharma/Nycomed, Zgierz
- South Africa (12):
  - Altana Pharma/Nycomed, Arcadia, Pretoria
  - Altana Pharma/Nycomed, Bellville, Cape Town
  - Altana Pharma/Nycomed, Cape Town
  - Altana Pharma/Nycomed, Cape Town, Tygerberg
  - Altana Pharma/Nycomed, Durbanville / Cape Town
  - Altana Pharma/Nycomed, Gatesville, Cape Town
  - Altana Pharma/Nycomed, Lyttleton
  - Altana Pharma/Nycomed, Mowbray, Cape Town
  - Altana Pharma/Nycomed, Observatory Cape
  - Altana Pharma/Nycomed, Pretoria
  - Altana Pharma/Nycomed, Westville
  - Altana Pharma/Nycomed, Wynberg

REFERENCES:
- See also: BY9010_M1-142 Synopsis.pdf — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=4523&filename=BY9010_M1-142%20Synopsis.pdf